CLINICAL TRIAL: NCT00144755
Title: Intensified CHOP Plus Rituximab (R-CHOP 14) Versus CHOP Plus Rituximab (R-CHOP 21) and Frontline/Prophylactic Darbepoetin Alfa Treatment Versus Usual Symptomatic Treatment of Anemia in Patients Aged 60 to 80 Years With Diffuse Large B-cell Lymphoma.
Brief Title: R-CHOP-14 Versus R-CHOP-21 and Darbepoetin Alpha in Patients Aged 60-80 Years With Diffuse Large B-cell Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lymphoma Study Association (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LNH03-6B
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Diffuse Large Cell Lymphoma
Keywords: lymphoma, diffuse large B-cell; rituximab; chemotherapy; erythropoetin; darbepoetin alfa
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- R-CHOP21 (Active Comparator): 8 cycles of R-CHOP21
  Interventions: Drug: Darbepoetin alfa
- R-CHOP21, Darbepoetin alfa (Experimental): 8 cycles of R-CHOP21 + prophylactic darbepoetin alfa
  Interventions: Drug: Darbepoetin alfa
- R-CHOP14 (Experimental): 8 cycles of R-CHOP14
  Interventions: Drug: Darbepoetin alfa
- R-CHOP14, Darbepoetin alfa (Experimental): 8 cycles of R-CHOP14 + prophylactic darbepoetin alfa
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Darbepoetin alfa — prophylactic administration of darbepoetin alfa in experimental arm

SUMMARY:
This study is a multicentric randomized trial evaluating the efficacy and safety of R-CHOP given every 14 days compared to R-CHOP given every 21 days in association or not with darbepoetin alfa in order to maintain hemoglobin above 13 g/dl, compared to classical symptomatic treatment of anemia in patients aged from 60 to 80 years with diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
In patients aged 60 to 75 years with diffuse large B-cell lymphoma, the shortening of interval between the courses of CHOP combination (CHOP-14), improves the complete response rate, the progression free survival and the overall survival.

The addition of Rituximab to standard CHOP (R-CHOP) has also been shown to improve complete remission rate (CR), event-free survival (EFS) and overall survival (OS) in elderly patients with B-DLCL.

The aim of this study is to test the hypothesis that the increase of the dose intensity by shortening the interval between two courses of R-CHOP (R-CHOP-14)could further improve the results of the R-CHOP.

Anemia is frequent at diagnosis and during the treatment of aggressive lymphoma. In the previous LNH 98-5 study, 72 % of the patients had, at the diagnosis, a hemoglobin level inferior to 13 g/dl. Moreover, during the treatment, 92 % of the patients had a hemoglobin level less than 13 g/dl and 30 % were transfused. The presence of anemia at diagnosis is an indicator of poor prognosis in multivariate analysis. This prognosis impact could probably be explained at cellular level on the tumor. Tumoral hypoxia is increased by the presence of anemia. Due to this hypoxia, the expression of tumor growth factor may be increased: e.a VEGF and the induction of expression of multi drug resistance (MDR1) is observed. This resistance to treatment is also due to the inhibition of genotoxic activity of free radicals induced by ionised radiation and chemotherapy. Experimentally, the negative impact of hypoxia on the efficacy of chemotherapy has been demonstrated in sarcoma cell lines for doxorubicin, vincristine and all most cyclophosphamide. Finally, hypoxia induced over expression of apoptosis resistance genes and induced a growth advantage for apoptosis resistant tumoral lines. Improvement of survival in patients receiving erythropoetin with chemotherapy or radiotherapy was suggested in a study on patients treated with a neoadjuvant radiochemotherapy for head and neck cancer. Erythropoetin could act to protect several normal tissues during chemotherapy and thus could decrease treatment related morbidity. Darbepoetin alfa is a new recombinant protein stimulating erythropoiesis. Thus, the use of darbepoetin alfa, in association with chemotherapy, could increase CR rate, EFS and OS in patients treated for diffuse large B-cell lymphoma.

This study is a multicentric, phase III open-label, randomized trial evaluating the efficacy and safety of R-CHOP given every 14 days compared to R-CHOP given every 21 days in association or not with darbepoetin alfa in order to maintain hemoglobin above 13 g/dl, compared to classical symptomatic treatment of anemia in patients aged 66 to 80 years with not previously treated diffuse large B-cell lymphoma with at least one adverse prognostic factor of the age adjusted IPI.

ELIGIBILITY:
Inclusion Criteria:

Patients with histologically proven CD20+ diffuse large B cell lymphoma (WHO Classification).

Aged 66 to 80 years old. Patients not previously treated. Ann Arbor stage II, III, IV. ECOG performance status 0 to 2. Age-adjusted IPI equal to 1, 2, or 3. With a minimum life expectancy of 3 months. Negative HIV, HBV and HCV serologies test < 4 weeks (except after vaccination for HBV).

Having signed a written informed consent.

Exclusion Criteria:

Any other histological type of lymphoma. Any history of treated or non-treated indolent lymphoma. However, patients not previously diagnosed and having a diffuse large B-cell lymphoma with some small cell infiltration in bone marrow or lymph node may be included.

Central nervous system or meningeal involvement by lymphoma. Contra-indication to any drug contained in the chemotherapy regimens. Any serious co-morbid active disease (according to the investigator's decision).

Poor renal function (creatinin level > 150 micromol/l), poor hepatic function (total bilirubin level > 30mmol/l, transaminases > 2.5 maximum normal level) unless these abnormalities are related to the lymphoma.

Poor bone marrow reserve as defined by neutrophils < 1.5 G/l or platelets < 100 G/l, unless related to bone marrow infiltration.

Any history of cancer during the last 5 years with the exception of non-melanoma skin tumors or stage 0 (in situ) cervical carcinoma.

Uncontrolled hypertension. Known hypersensitivity to erythropoietin. Myocardial infarction during last 3 month, or unstable coronary disease, or uncontrolled cardiac insufficiency.

Venous thrombosis or pulmonary embolism during last 3 months. Treatment with any investigational drug within 30 days before planned first cycle of chemotherapy and during the study.

Pregnant or lactating women. Adult patient under tutelage.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2003-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of R-CHOP 14 vs R-CHOP 21 measured by event-free survival (EFS) | 8 years

SECONDARY OUTCOMES:
Efficacy of darbepoetin alfa in association with chemotherapy measured by the EFS. | 8 years
Efficacy and toxicity of R-CHOP 14 vs R-CHOP 21 | 8 years
  CR rate, DFS, OS, dose intensity and additional toxicities.
Efficacy and toxicity of Darbepoetin alfa in association with R-CHOP. | 8 years
  event-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Richard Delarue, MD, Principal Investigator — Lymphoma Study Association; André Bosly, MD, Study Director — Lymphoma Study Association; Corinne Haioun, MD, Study Chair — Lymphoma Study Association; Hervé Tilly, MD, Study Chair — Lymphoma Study Association
Locations (14):
- Belgium (2):
  - Université de Gent, Ghent
  - Groupe d'Etude des Lymphomes de l'adulte, Mont-Godinne
- France (11):
  - Polyclinique Bordeaux Nord, Bordeaux
  - Hôpital Henri Mondor, Créteil
  - Hématologie CHU de Lille, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital Saint Louis, Paris
  - Hématologie Adultes - Hôpital Necker, Paris
  - Service d'Hématologie - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Centre Hospitalier Robert Debré, Reims
  - Centre Henri Becquerel, Rouen
  - Hématologie CHU Purpan, Toulouse
  - Institut Gustave Roussy, Villejuif
- Schweirische Arbeitsgruppe fur klinische Krebsforschung, Lausanne, Switzerland

REFERENCES:
- [Background] Feugier P, Van Hoof A, Sebban C, Solal-Celigny P, Bouabdallah R, Ferme C, Christian B, Lepage E, Tilly H, Morschhauser F, Gaulard P, Salles G, Bosly A, Gisselbrecht C, Reyes F, Coiffier B. Long-term results of the R-CHOP study in the treatment of elderly patients with diffuse large B-cell lymphoma: a study by the Groupe d'Etude des Lymphomes de l'Adulte. J Clin Oncol. 2005 Jun 20;23(18):4117-26. doi: 10.1200/JCO.2005.09.131. Epub 2005 May 2. PMID 15867204
- [Background] Pfreundschuh M, Trumper L, Kloess M, Schmits R, Feller AC, Rube C, Rudolph C, Reiser M, Hossfeld DK, Eimermacher H, Hasenclever D, Schmitz N, Loeffler M; German High-Grade Non-Hodgkin's Lymphoma Study Group. Two-weekly or 3-weekly CHOP chemotherapy with or without etoposide for the treatment of elderly patients with aggressive lymphomas: results of the NHL-B2 trial of the DSHNHL. Blood. 2004 Aug 1;104(3):634-41. doi: 10.1182/blood-2003-06-2095. Epub 2004 Mar 11. PMID 15016643
- [Derived] Camus V, Belot A, Oberic L, Sibon D, Ghesquieres H, Thieblemont C, Fruchart C, Casasnovas O, Michot JM, Molina TJ, Bosly A, Joubert C, Haioun C, Nicolas-Virelizier E, Feugier P, Fitoussi O, Delarue R, Tilly H. Outcomes of older patients with diffuse large B-cell lymphoma treated with R-CHOP: 10-year follow-up of the LNH03-6B trial. Blood Adv. 2022 Dec 27;6(24):6169-6179. doi: 10.1182/bloodadvances.2022007609. PMID 35737565
- [Derived] Petrella T, Copie-Bergman C, Briere J, Delarue R, Jardin F, Ruminy P, Thieblemont C, Figeac M, Canioni D, Feugier P, Fabiani B, Leroy K, Parrens M, Andre M, Haioun C, Salles GA, Gaulard P, Tilly H, Jais JP, Molina TJ. BCL2 expression but not MYC and BCL2 coexpression predicts survival in elderly patients with diffuse large B-cell lymphoma independently of cell of origin in the phase 3 LNH03-6B trial. Ann Oncol. 2017 May 1;28(5):1042-1049. doi: 10.1093/annonc/mdx022. PMID 28327893
- [Derived] Ghesquieres H, Larrabee BR, Haioun C, Link BK, Verney A, Slager SL, Ketterer N, Ansell SM, Delarue R, Maurer MJ, Fitoussi O, Habermann TM, Peyrade F, Dogan A, Molina TJ, Novak AJ, Tilly H, Cerhan JR, Salles G. FCGR3A/2A polymorphisms and diffuse large B-cell lymphoma outcome treated with immunochemotherapy: a meta-analysis on 1134 patients from two prospective cohorts. Hematol Oncol. 2017 Dec;35(4):447-455. doi: 10.1002/hon.2305. Epub 2016 Jun 10. PMID 27282998
- [Derived] Copie-Bergman C, Cuilliere-Dartigues P, Baia M, Briere J, Delarue R, Canioni D, Salles G, Parrens M, Belhadj K, Fabiani B, Recher C, Petrella T, Ketterer N, Peyrade F, Haioun C, Nagel I, Siebert R, Jardin F, Leroy K, Jais JP, Tilly H, Molina TJ, Gaulard P. MYC-IG rearrangements are negative predictors of survival in DLBCL patients treated with immunochemotherapy: a GELA/LYSA study. Blood. 2015 Nov 26;126(22):2466-74. doi: 10.1182/blood-2015-05-647602. Epub 2015 Sep 15. PMID 26373676
- [Derived] Delarue R, Tilly H, Mounier N, Petrella T, Salles G, Thieblemont C, Bologna S, Ghesquieres H, Hacini M, Fruchart C, Ysebaert L, Ferme C, Casasnovas O, Van Hoof A, Thyss A, Delmer A, Fitoussi O, Molina TJ, Haioun C, Bosly A. Dose-dense rituximab-CHOP compared with standard rituximab-CHOP in elderly patients with diffuse large B-cell lymphoma (the LNH03-6B study): a randomised phase 3 trial. Lancet Oncol. 2013 May;14(6):525-33. doi: 10.1016/S1470-2045(13)70122-0. Epub 2013 Apr 9. PMID 23578722
- See also: Official site of the Groupe d'Etudes des Lymphomes de l'Adulte (In french) — http://www.gela.org